CLINICAL TRIAL: NCT04647942
Title: Is Meniscal Volume Critical to Post-meniscectomy Symptoms? A Retrospective Study
Brief Title: Is Meniscal Volume Critical to Post-meniscectomy Symptoms?
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: V1 07112013
Record Dates: First submitted 2013-12-22; First posted 2020-12-01 (Actual); Last update posted 2020-12-01 (Actual); Status verified 2020-11

CONDITIONS: Meniscal Tear
Keywords: meniscectomy; volume; pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Meniscectomy: Patients who underwent a meniscectomy

SUMMARY:
With this study we would like to investigate whether a certain, critical loss of meniscal volume, is critical to the development of pain.

DETAILED DESCRIPTION:
1. Background and rationale It is known that a partial meniscectomy of the knee is a risk factor to the development of early osteoarthritis with complaints of pain.
2. Trial objectives and Design 2.1 Trial objectives With this study we would like to investigate whether a certain, critical loss of meniscal volume, is critical to the development of pain.

   2.2 Primary endpoints How much volume can be resected peroperatively without developing postoperative pain.

   2.3 Secondary endpoints A possible correlation between the resected volume and the severity of the pain.
3. Selection and withdrawal of subjects

3.1 Inclusion criteria

* All patients who were treated with a partial meniscectomy for a meniscal tear and have postoperative MRI's.
* Age between 14 and 50 years old
* Women of child bearing age can be included: the study has no effect on their methods of contraception.

3.2 Exclusion criteria

* A history of a tibia plateau fracture or severe deformity of the knee
* Rupture of the ACL/PCL/collateral ligaments of the knee
* Focal cartilage defects of the knee

ELIGIBILITY:
Inclusion Criteria:

* All patients who were treated with a partial meniscectomy for a meniscal tear and have postoperative MRI's.
* Age between 14 and 60 years old
* Women of child bearing age can be included: the study has no effect on their methods of contraception.

Exclusion Criteria:

* A history of a tibia plateau fracture or severe deformity of the knee
* Rupture of the ACL/PCL/collateral ligaments of the knee
* Focal cartilage defects of the knee

Ages: 14 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: * All patients who were treated with a partial meniscectomy for a meniscal tear and have postoperative MRI's.
  * Age between 14 and 60 years old
  * Women of child bearing age can be included: the study has no effect on their methods of contraception.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
How much volume can be resected peroperatively without developing postoperative pain. | 3 years
  A possible correlation between the resected volume and the severity of the pain.

CONTACTS AND LOCATIONS:
Overall Officials: Johan Bellemans, MD, PhD, Study Director — UZ Leuven
Locations (1):
- University Hospitals of Leuven, Leuven, Antwerp, Belgium